CLINICAL TRIAL: NCT05349474
Title: A Double-blind, Placebo Controlled Trial of Metformin Treatment in Progressive Multiple Sclerosis
Brief Title: Metformin Treatment in Progressive Multiple Sclerosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kevin Patel, Assistant Professor, Department of Neurology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-000020
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Secondary Progressive Multiple Sclerosis; Primary Progressive Multiple Sclerosis
Keywords: Multiple sclerosis; Demyelinating disease
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Demyelinating Diseases | interventions — Metformin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin Treatment (Experimental): Metformin 500 mg tablets up to 2,000 mg (4 tablets) a day divided into two doses. Patients will start on 500 mg Qday and a titration to maximum dose will be attempted during the first 30 day period of the study.
  Interventions: Drug: Metformin 500 Mg Oral Tablet, up to 4 tablets a day
- Placebo Treatment (Placebo Comparator): Placebo tablets identical to metformin 500 mg tablets divided into two doses. Patients will be started on 1 tablet a day and a titration to maximum dose (4 tablets) will be attempted during the first 30 day period of the study.
  Interventions: Drug: Placebo oral tablet identical to metformin, up to 4 tablets a day

INTERVENTIONS:
Drug: Metformin 500 Mg Oral Tablet, up to 4 tablets a day — Metformin 500 mg oral tablets to be titrated to 2000 mg/day divided over two doses or maximum tolerated dose
  Arms: Metformin Treatment
Drug: Placebo oral tablet identical to metformin, up to 4 tablets a day — Placebo tablets identical to metformin tablets. To be titrated to four tablets divded over two doses or maximum tolerated dose
  Arms: Placebo Treatment

SUMMARY:
The purpose of this study is to assess the safety of metformin for treatment of progressive multiple sclerosis

DETAILED DESCRIPTION:
This will be a single site 1:1 randomized, placebo controlled trial of metformin treatment vs matching placebo in 44 men and women with primary progressive multiple sclerosis and secondary multiple sclerosis, without diabetes, not treated with metformin aged 30-65. The trial will last 12 months and have 3 study visits, baseline, 6 months, and 12 months. The trial will be preceded by a screening period. Over the initial 30 day titration period subjects will be titrated from 500 mg a day to 2,000 mg of metformin in increments of 500 mg every 10 days. Patients will remain on their tolerated dose and included in analysis on an intent to treat basis. Brain MRI, cognitive testing and clinical measures will be collected at baseline, month 6 and month 12. OCT will be collected at baseline and month 12. The primary outcomes are the following safety outcomes: 1) number of patients with adverse events 2) number of patients with laboratory abnormalities 3) number of patients with new T2 lesions on MRI. The secondary outcomes include reduction in localized cortical thinning on brain MRI; reduction in thalamic atrophy on brain MRI. Further exploratory outcomes include 1) improvement in SDMT-oral score, 2) improvement in CVLT-II score, 3) improvement in PACC score 4) improvement in PASAT score. Exploratory outcomes include 1) Decrease in plasma neurofilament light chain levels, 2) Reginal nerve fiber layer preservation on OCT, 3) Ganglion cell inner plexiform layer preservation, and 4) Percentage of phase rim lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patient signed informed consent.
2. Age 30-65
3. Primary Progressive Multiple Sclerosis or Secondary Progressive Multiple Sclerosis as defined by the 2017 McDonald Criteria
4. Intent to maintain current MS disease modifying treatment through the trial duration

Exclusion Criteria:

1. Clinical relapse in prior 12 months
2. New T2 lesion or gadolinium enhancing lesion in prior 12 months
3. Glucocorticoid use in prior six months outside the context of premedication for disease modifying treatment
4. Changes in disease modifying therapy in prior three months
5. Plans to change current disease modifying therapy
6. Contraindication to MRI, inability to tolerate MRI
7. Use of metformin for any other indication
8. Renal dysfunction (GFR < 60)
9. Hepatic dysfunction (AST or ALT > 1.5 x upper limit of normal)
10. B12 deficiency
11. Prior poor reaction to metformin
12. Congestive heart failure
13. Alcohol abuse
14. Metabolic acidosis
15. Females who are pregnant or who plan to become pregnant during the 12 months of enrollment, or who wish to breastfeed during any part of the 12 months of enrollment
16. Concomitant use of drugs with drug-drug interactions with metformin
17. Previous adverse effect with metformin treatment

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
number of patients with adverse events between baseline and conclusion (month 0 and month 12) | between month 0 and month 12
  number of patients with adverse events comparing the two treatment groups
number of patients with laboratory abnormalities between baseline and conclusion (month 0 and month 12) | between month 0 and month 12
  number of patients with laboratory abnormalities comparing the two treatment groups
number of patients with new T2 lesions on MRI from baseline to conclusion (month 0 and month 12) | between month 0 and month 12
  number of patients with new T2 lesions comparing the two treatment groups

SECONDARY OUTCOMES:
a reduction in localized cortical thinning on brain MRI between baseline and conclusion (month 0 and month 12) | between month 0 and month 12
  a reduction in localized cortical thinning on brain MRI comparing the two treatment groups
a reduction in thalamic atrophy on brain MRI between baseline and conclusion (month 0 and month 12) | between month 0 and month 12
  a reduction in thalamic atrophy on brain MRI comparing the two treatment groups

OTHER OUTCOMES:
improvement in SDMT-oral score between baseline and conclusion (month 0 and month 12) | between month 0 and month 12
  improvement in SDMT-oral score between comparing the two treatment groups
improvement in CVLT-II score between baseline and conclusion (month 0 and month 12) | between month 0 and month 12
  improvement in CVLT-II score between comparing the two treatment groups
improvement in PACC score between baseline and conclusion (month 0 and month 12) | between month 0 and month 12
  improvement in PACC score between comparing the two treatment groups
improvement in PASAT score between baseline and conclusion (month 0 and month 12) | between month 0 and month 12
  improvement in PASAT score between comparing the two treatment groups
decrease in plasma neurofilament light chain levels between baseline and conclusion (month 0 and month 12) | between month 0 and month 12
  decrease in plasma neurofilament light chain levels comparing the two treatment groups
decrease in number of phase rimmed lesions between baseline and conclusion (month 0 and month 12) | between month 0 and month 12
  decrease in number of phase rimmed lesions comparing the two treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Patel, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No